CLINICAL TRIAL: NCT04659538
Title: A Prospective, Single Arm, FIH Study to Evaluate the Safety and Feasibility of the CAPTIS Device in Patients Undergoing Transcatheter Aortic Valve Replacement (TAVR)
Brief Title: The CAPTIS® Study - Embolic Protection in TAVR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Filterlex Medical Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: CLD-FLX-001
Record Dates: First submitted 2020-11-17; First posted 2020-12-09 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAPTIS Embolic Protection (Experimental): TAVR will be performed according to standard institutional practice under local or general anesthesia by the transfemoral approach. The investigational device will be advanced and deployed across the aortic arch covering the ostia of the 3 great vessels (innominate, left carotid, and left-subclavian arteries) at the initiation of the procedure and withdrawn at the completion of the TAVR procedure.
  Interventions: Device: CAPTIS Embolic Protection device

INTERVENTIONS:
Device: CAPTIS Embolic Protection device — The CAPTIS Embolic Protection device will be deployed during standard of care TAVR procedure. The device's safety will be assessed up to one month post procedure. The device's technical performance and feasibility to capture and remove debris during the procedure will be evaluated.

SUMMARY:
This is a First in Human study with the Filerlex CAPTIS device designed to demonstrate the safety and feasibility of the device in subjects undergoing Transcatheter Aortic Valve Replacement (TAVR)

DETAILED DESCRIPTION:
This is a prospective, multi center, single arm, FIH safety and feasibility study enrolling up to 20 patients. Patients undergoing clinically indicated TAVR who comply with the study inclusion/exclusion criteria will be enrolled to have embolic protection with the CAPTIS® Device during the TAVR procedure.

Screening activities will include initial screening by the site, analysis of patient CT scan by the sponsor and core-lab, and review of the clinical and imaging data by an eligibility committee to confirm that all inclusion/exclusion criteria are met. Final eligibility for study enrollment is then determined by the investigator in the cardiac catheterization laboratory.

Enrolled patients will undergo safety assessment during the procedure, post-procedure, and at 30 days post-procedure; Feasibility evaluation will be assessed during procedure.

ELIGIBILITY:
Inclusion Criteria:

1. The patient must be ≥18 years of age.
2. Patient has clinical indications for TAVR procedure.
3. TAVR procedure planned with femoral artery access site
4. TAVR device approved for use in the US, Europe or Israel
5. Femoral and iliac artery with a minimal luminal diameter of at least 6 mm
6. Descending Aorta diameter of 20 to 27mm measured 10cm from the left subclavian, determined by CT scan analysis
7. The distance between the innominate and left-subclavian arteries (including their lumens) is less than 65mm
8. Patient is willing to comply with protocol-specified preprocedure and follow-up evaluations.
9. The patient has been informed of the nature of the trial, agrees to its provisions and has provided written informed consent as approved by the ethics committee of the clinical site.

Exclusion Criteria:

General

1. Pregnant or nursing female patients. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to surgical procedure per site standard test
2. Hemodialysis shunt, graft, or arterio-venous fistula involving the lower extremity vasculature
3. Blood dyscrasias: WBC <5000/microliter, Hb <10.0 mg/dL, PLT <100,000/microliter, history of bleeding diathesis, coagulopathy, or conditions associated with increased thrombogenicity
4. Hemodynamic instability requiring pharmacological or mechanical circulatory support. Patient in whom hemodynamic instability is expected or at increased risk, will also be excluded.
5. Any surgery or procedure (including endovascular) planned for the 30 days post TAVR
6. Severe left-ventricle dysfunction with LVEF ≤30%
7. Echocardiographic evidence of intracardiac or aortic mass, thrombus, or vegetation
8. Active or recent bacterial endocarditis
9. Active peptic ulcer or upper GI bleeding within the prior 3 months
10. A known hypersensitivity or contraindication to aspirin, heparin, bivalirudin, clopidogrel, ticagrelor, or contrast media, which cannot be adequately pre-medicated or replaced by an alternative agent
11. Renal insufficiency (GFR < 30). Patients on renal replacement therapy (dialysis) can be enrolled into the study.
12. Life expectancy < 12 months due to non-cardiac comorbid conditions
13. Patients who refuse blood transfusion
14. Chronic or persistent atrial fibrillation, frequent recurring atrial fibrillation, and patients with planned ablation for atrial fibrillation
15. Currently participating in another investigational drug or device study
16. Patient is otherwise not appropriate for the study as determined by the investigator or the Eligibility Committee

    Neurologic
17. Prior CVA or a TIA
18. Patient has undergone carotid stenting or carotid endarterectomy within the previous 6 months
19. Patient has active major psychiatric disease that prevent a conscious consent
20. Patient with neurodegenerative or other progressive neurological disease or history of significant head trauma followed by persistent neurologic deficit or known structural brain abnormalities

    Vascular
21. Severe tortuosity or luminal diameter of less than 6 mm of the femoral or iliac arteries
22. Excessive tortuosity or calcification or atherosclerosis of any segment of the aorta and iliac arteries
23. Patient whose innominate, carotid, or subclavian arteries reveals significant stenosis, ostial calcification, ectasia, dissection, or aneurysm at the ostium

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-24 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-05-03 (Actual)

PRIMARY OUTCOMES:
Safety - Occurrence of MACCE | 72 hours
  Occurrence of all MACCE at 72 hours post procedure, with MACCE defined as all death and all cerebrovascular events (all TIA and stroke).
Safety - Device related complications | 72 hours
  Number of device related complications [at 72 hours]

SECONDARY OUTCOMES:
Secondary Safety - Occurrence of MACCE | 30 days
  All MACCE, number of stroke events, number of TIA events [at 30 days]
Secondary Safety - Acute Kidney Injury | 72 hours
  Number of subjects with acute kidney injury (defined as increase in creatinine level of 25% or 0.5mg/dL at 72 hours (or discharge) as compared to pre-procedure baseline)
Device feasibility - Histopathologic examination of debris captured and removed by the device | Day 0
  All devices will be sent for histopathologic examination to determine the device's feasibility to catch and remove debris during the TAVR procedure
Technical Device Performance - the ability to deploy and retrieve the device without device malfunction | Day 0
  Number of procedures performed without device malfunction

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (3):
  - Wolfson Medical Center, Holon
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Sponsor website — http://filterlex.com